CLINICAL TRIAL: NCT02793154
Title: A Randomized, Open-label, Active-Controlled, Parallel-Group, Exploratory Study on the Effects of Repeated Doses of Albiglutide Compared to Exenatide on Gastric Myoelectrical Activity and Gastric Emptying in Subjects With Type 2 Diabetes Mellitus
Brief Title: An Exploratory Study on the Effects of Repeat Doses of Albiglutide Compared to Exenatide on Gastric Myoelectrical Activity and Gastric Emptying in Type 2 Diabetes Mellitus Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination due to insufficient enrollment.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Wake Forrest Baptist Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204879
Record Dates: First submitted 2016-05-16; First posted 2016-06-08 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: gastric emptying; albiglutide; GMA; exenatide; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; rGLP-1 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: Exenatide (Experimental): Part A is a single arm design and all subjects will receive 10 mcg subcutaneous injection (SC) of exenatide twice daily for 5 days
  Interventions: Drug: Exenatide
- Part B: Albiglutide (Experimental): In Part B, half of the subjects will be randomized to receive albiglutide: On Day 1: Once weekly SC injection at 30 mg for 4 weeks From Week 5, Day 1: Dose will be increased to 50 mg once weekly SC injection for 4 weeks
  Interventions: Drug: Albiglutide
- Part B: Exenatide (Active Comparator): In Part B, half of the subjects will be randomized to receive exenatide: On Day 1: Twice daily SC injection at 5 mcg for 4 weeks.
  From Week 5, Day 1: Dose will be uptitrated to 10 mcg twice daily SC injection for 4 weeks
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Supplied as SC injection containing 250 mcg/mL of exenatide, provided in the following dose regimens: Part A: 10 mcg taken twice daily for 5 days; Part B: 5 mcg twice daily taken for 4 weeks followed by uptitration to 10 mcg for 4 weeks In both parts, it will be administered within 60-minute period before morning and evening meals (or before 2 meals with approximate >=6 hours apart)
  Other Names: Byetta
  Arms: Part A: Exenatide; Part B: Exenatide
Drug: Albiglutide — Part B: Albiglutide will be supplied as follows:30 mg SC injection pen containing 40.3 mg lyophilized albiglutide and 0.65 mL; 50 mg SC injection pen contains 67 mg lyophilized albiglutide and 0.65 mL water; Starting dose will be 30 mg weekly for 4 weeks and then uptitrated to 50 mg weekly for 4 weeks; Administered as a single SC injection once a week in the morning
  Other Names: Tanzeum in US
  Arms: Part B: Albiglutide

SUMMARY:
The primary objective of this study is to compare the effect of albiglutide and exenatide on gastric myoelectrical activity (GMA), gastric emptying (GE) and nausea (as measured by visual analogue scale [VAS]) in subjects with type 2 diabetes mellitus (T2DM). The study is divided in two parts. Part A will characterize the GMA, GE and nausea response to exenatide and confirm exenatide as a positive control for Part B. Part B will compare the effects of albiglutide and exenatide on GMA, GE and nausea.

Part A is a single arm, open-label design and all subjects will receive 10 microgram (mcg) subcutaneous exenatide twice daily for 5 days. This part will comprise 3 study periods: a 3-week screening/wash-out, 5-day treatment, and follow-up (within 7 days after the last dose of exenatide). The total duration of a subject's participation in Part A will be approximately 5 weeks. Once Part A is complete, data will be reviewed and a decision to progress to Part B will be made.

In Part B, subjects will be randomized 1:1 to receive either albiglutide (starting dose of 30 milligrams [mg] once weekly for 4 weeks, followed by 50 mg once weekly for 4 weeks) or exenatide (starting dose of 5 mcg twice daily for 4 weeks, followed by 10 mcg twice daily for 4 weeks). The total duration of a subject's participation in the study will be approximately 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 and 60 years of age at the time of signing the informed consent.
* Type 2 diabetes mellitus diagnosed at least 6 months prior to screening.
* Subjects treated with diet and exercise alone or stable dose of single oral antihyperglycemic medication (OAM) of metformin, sulfonylurea (except chlorpropamide), sodium glucose co-transporter 2-inhibitor, or meglitinide for at least 2 months prior to screening
* Glycated hemoglobin A1C (HbA1c) >6.5% and <=9.0% at screening. If the first HbA1c value does not meet eligibility criterion, the HbA1c may be rechecked once during screening. If the average of these determinations meets the criterion, the subject is eligible.
* Fasting plasma glucose (FPG) <=210 mg/deciliter (dL; central lab) at screening. If the first FPG value does not meet eligibility criterion, the FPG may be rechecked once during screening.
* Patient assessment of upper GI symptom severity index at screening:

Overall score <=20 (if score is >=21 and <=25, subjects can be re-evaluated 2 weeks later) Total score of items 1-9 is <=9 Score from any of single item <=2

* Body mass index (BMI) >20 kilograms (kg)/meter (m)^2 and <35 kg/m^2 and a stable weight (no more than 5% reported change within 3 months prior to screening).
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test for females of reproductive potential [FRP] only), not breastfeeding, and at least one of the following conditions applies:

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP (eg., combined oral contraceptive pill) from 30 days prior to the first dose of study medication and until after the last dose of study medication and completion of the follow-up visit.

Non-reproductive potential defined as either:

* Pre-menopausal with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; or documented bilateral oophorectomy, or;
* Postmenopausal defined as 12 months of spontaneous amenorrhea and age appropriate (i.e., >50 years). In questionable cases, a blood sample with simultaneous follicle stimulating hormone >40 milli-International units/milliliters (mL) and estradiol <40 picograms/mL (<140 picomoles/L) is confirmatory, depending on local laboratory ranges. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment

  * For the regular use of other medications (does not include protocol excluded medications), subjects must be on a stable dose for at least 4 weeks before screening
  * Capable of giving signed informed consent; which includes compliance with the requirements and restrictions listed in the consent form and in this protocol

Exclusion Criteria:

* Type 1 diabetes mellitus
* Type 2 diabetes mellitus treated with more than one OAM or with chronic use of insulin within 3 months prior to screening
* Hemoglobin <11 grams (g)/dL (<110 g/L) for male subjects and <10 g/dL (<100 g/L) for female subjects at screening
* Fasting triglyceride level >500 mg/dL at screening
* Hemoglobinopathy that may affect proper interpretation of HbA1c
* History of cancer that has not been in full remission for at least 3 years before screening. (A history of squamous cell or basal cell carcinoma of the skin or treated cervical intra-epithelial neoplasia I or II is allowed).
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* History of acute or chronic pancreatitis.
* History or current severe lactose intolerance
* History of thyroid dysfunction or an abnormal (i.e., outside the normal reference range) thyroid function test assessed by thyroid stimulating hormone at screening.
* Alanine aminotransferase (ALT) >2.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Clinical diagnosis of gastroparesis.
* History of significant GI medical conditions such as chronic esophagitis, peptic ulcer diseases, celiac disease, inflammatory bowel disease, unexplained abdominal pain or irritable bowel syndrome and/or history of surgery that in the opinion of the investigator is likely to significantly affect upper GI or pancreatic function (e.g., gastric bypass, gastric banding, antrectomy, Roux en Y bypass, gastric vagotomy, small bowel resection, or surgeries thought to significantly affect upper GI function).
* History of hypoglycemia unawareness (i.e., the absence of autonomic warning symptoms before the development of neuroglycopenic symptoms such as blurred vision, difficulty speaking, feeling faint, difficulty thinking, and confusion).
* Diabetic complications (e.g., active proliferative retinopathy or severe diabetic neuropathy) or any other clinically significant abnormality (including a psychiatric disorder) that, in the opinion of the investigator, may pose additional risk in administering the investigational product or may influence data interpretation.
* Clinically significant cardiovascular and/or cerebrovascular disease at any time, such as prior myocardial infarction, unstable angina, stroke, transient ischemic attack or documented heart failure, before screening.
* Estimated glomerular filtration rate (eGFR) <=75 mL/min/1.73 m^2 (calculated using the MDRD formula) at screening.
* Lung diseases associated with pulmonary dysfunction (e.g. chronic obstructive pulmonary disease).
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied should be excluded unless the investigator (in consultation with the Medical Monitor, if necessary) decides and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or ability to interpret study results
* Unable to refrain from medications that might modify GMA or GI motility, such as prokinetics (e.g., erythromycin), anti-emetics (e.g., metoclopromide), narcotics (e.g., morphine), anticholinergics (e.g.,domperidone), anti-acids (e.g., proton pump inhibitors, H2 blockers) and laxatives, received within 7 days prior to screening or high likelihood of a requirement during the study.
* Use of oral or systemically injected glucocorticoids within the 3 months prior to randomization or high likelihood of a requirement for prolonged treatment (>1 week) in the 4months following randomization. However, short courses of oral steroids (single dose or multiple doses for up to 7 days) may be permitted provided these cases are discussed with the Medical Monitor. Inhaled, intra-articular, epidural, and topical corticosteroids are allowed
* Known allergy to albiglutide, exenatide or any product components (including yeast and human albumin), any other glucagon-like receptor 1 analogue, or other study treatment excipients OR other contraindications (per the principal investigator) for the use of potential study treatment.
* Intolerance or allergy to any component of GE test meal
* Received any glucagon-like peptide 1 receptor agonist at any time
* Receipt of any investigational drug within the 30 days or 5 half-lives, whichever is longer, before screening, a history of receipt of an investigational antidiabetic drug within the 3 months before randomization.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study compared effects of repeated doses of albiglutide and exenatide in type 2 diabetes mellitus. This study was conducted in two parts; first cohort of participants (Par.) were planned to receive exenatide (Part A) and second cohort with albiglutide or exenatide (Part B). There were no pre-specified Primary or Secondary endpoints for Part A.
Pre-assignment Details: This study was terminated during exploratory Part A due to the difficulty with enrollment and Part B was cancelled. Hence, Par. received only exenatide subcutaneous (SC) injection in Part A. The data was only collected in Part A and no Par. were enrolled in Part B. All the 4 enrolled Par. completed Part A and no Par. was withdrawn from study.
Groups:
- Part A: Exenatide SC Injection: Eligible Par. received 10 micrograms of exenatide twice daily for 5 days injected subcutaneously into in the abdomen, thigh or upper arm region using a prefilled injector pen. Exenatide was administered via an auto-injector within 60 minutes before the morning and evening meals.
- Part B: Exenatide SC Injection: Eligible Par. were planned to receive 5 micrograms of exenatide twice daily for 4 weeks, then up-titrated to 10 micrograms twice daily for 4 weeks injected subcutaneously into the abdomen, thigh or upper arm region using a prefilled injector pen. Exenatide was to be administered via an auto-injector within 60 minutes before the morning and evening meals.
- Part B: Albiglutide SC Injection: Eligible Par. were planned to receive 30 milligrams of albiglutide, weekly for 4 weeks, then up titrated to 50 milligrams, weekly for 4 weeks injected subcutaneously into the abdomen, thigh or upper arm region using a prefilled injector pen in the morning.
Period: Part A (Single Group-up to 12 Days)
Arm/Group | Part A: Exenatide SC Injection | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Started | 4 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B (Parallel Group-up to 84 Days)
Arm/Group | Part A: Exenatide SC Injection | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part B was cancelled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Exenatide SC Injection | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (3.30) |  |  | 56.8 (3.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 3 |  |  | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 2 |  |  | 2
  White-White/Causasian/European Heritage | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A: Distribution of Average Power by Frequency Region
Description: The effect of exenatide on gastric myoelectrical activity was assessed by electrogastrogram (EGG) using water load test (WLT). EGG with WLT is a standardized test to induce gastric distention and measure myoelectrical responses. The gastric myoelectrical activity is generated by the pacemaker interstitial cells at a normal frequency of 3 cycles per minute. The shift of frequency from normal gastric myoelectrical activity to a slower rhythm is bradygastria or faster rhythm is tachygastria. Individual Par. data for distribution of average power in the bradygastria, normal, tachygastria and duodenal range during pre-WL and 10, 20 and 30 minutes post-WL after treatment with exenatide has been presented. The analysis was performed on Pharmacodynamic Population, which included all Par. who received at least one dose of study medication and had valid data.
Time Frame: Up to Day 4
Population: Pharmacodynamic Population
Measure: Number; unit: Percentage of power
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Percentage of power
  Par. 1; Day 1; Pre-WL; Bradygastria | 56.15
  Par. 1; Day 1; Pre-WL; Normal | 23.49
  Par. 1; Day 1; Pre-WL; Tachygastria | 17
  Par. 1; Day 1; Pre-WL; Duodenal | 3.35
  Par. 1; Day 1; 10 minutes Post-WL; Bradygastria | 93.97
  Par. 1; Day 1; 10 minutes Post-WL; Normal | 2.9
  Par. 1; Day 1; 10 minutes Post-WL; Tachygastria | 2.4
  Par. 1; Day 1; 10 minutes Post-WL; Duodenal | 0.73
  Par. 1; Day 1; 20 minutes Post-WL; Bradygastria | 57.13
  Par. 1; Day 1; 20 minutes Post-WL; Normal | 23.29
  Par. 1; Day 1; 20 minutes Post-WL; Tachygastria | 13.17
  Par. 1; Day 1; 20 minutes Post-WL; Duodenal | 6.41
  Par. 1; Day 1; 30 minutes Post-WL; Bradygastria | 43.44
  Par. 1; Day 1; 30 minutes Post-WL; Normal | 36.16
  Par. 1; Day 1; 30 minutes Post-WL; Tachygastria | 17.78
  Par. 1; Day 1; 30 minutes Post-WL; Duodenal | 2.62
  Par. 1; Day 4; Pre-WL; Bradygastria | 71.94
  Par. 1; Day 4; Pre-WL; Normal | 13
  Par. 1; Day 4; Pre-WL; Tachygastria | 9.51
  Par. 1; Day 4; Pre-WL; Duodenal | 5.55
  Par. 1; Day 4; 10 minutes Post-WL; Bradygastria | 43.99
  Par. 1; Day 4; 10 minutes Post-WL; Normal | 12.94
  Par. 1; Day 4; 10 minutes Post-WL; Tachygastria | 28.33
  Par. 1; Day 4; 10 minutes Post-WL; Duodenal | 14.74
  Par. 1; Day 4; 20 minutes Post-WL; Bradygastria | 73.87
  Par. 1; Day 4; 20 minutes Post-WL; Normal | 10.97
  Par. 1; Day 4; 20 minutes Post-WL; Tachygastria | 8.77
  Par. 1; Day 4; 20 minutes Post-WL; Duodenal | 6.39
  Par. 1; Day 4; 30 minutes Post-WL; Bradygastria | 48.87
  Par. 1; Day 4; 30 minutes Post-WL; Normal | 16.66
  Par. 1; Day 4; 30 minutes Post-WL; Tachygastria | 23.16
  Par. 1; Day 4; 30 minutes Post-WL; Duodenal | 11.31
  Par. 2; Day 1; Pre-WL; Bradygastria | 67.44
  Par. 2; Day 1; Pre-WL; Normal | 10.67
  Par. 2; Day 1; Pre-WL; Tachygastria | 17.2
  Par. 2; Day 1; Pre-WL; Duodenal | 4.68
  Par. 2; Day 1; 10 minutes Post-WL; Bradygastria | 94.05
  Par. 2; Day 1; 10 minutes Post-WL; Normal | 2.46
  Par. 2; Day 1; 10 minutes Post-WL; Tachygastria | 2.83
  Par. 2; Day 1; 10 minutes Post-WL; Duodenal | 0.67
  Par. 2; Day 1; 20 minutes Post-WL; Bradygastria | 85.64
  Par. 2; Day 1; 20 minutes Post-WL; Normal | 11.72
  Par. 2; Day 1; 20 minutes Post-WL; Tachygastria | 2.43
  Par. 2; Day 1; 20 minutes Post-WL; Duodenal | 0.22
  Par. 2; Day 1; 30 minutes Post-WL; Bradygastria | 77.34
  Par. 2; Day 1; 30 minutes Post-WL; Normal | 15.57
  Par. 2; Day 1; 30 minutes Post-WL; Tachygastria | 6.23
  Par. 2; Day 1; 30 minutes Post-WL; Duodenal | 0.86
  Par. 2; Day 4; Pre-WL; Bradygastria | 43.32
  Par. 2; Day 4; Pre-WL; Normal | 23.82
  Par. 2; Day 4; Pre-WL; Tachygastria | 18.71
  Par. 2; Day 4; Pre-WL; Duodenal | 14.14
  Par. 2; Day 4; 10 minutes Post-WL; Bradygastria | 84.23
  Par. 2; Day 4; 10 minutes Post-WL; Normal | 7.93
  Par. 2; Day 4; 10 minutes Post-WL; Tachygastria | 6.81
  Par. 2; Day 4; 10 minutes Post-WL; Duodenal | 1.02
  Par. 2; Day 4; 20 minutes Post-WL; Bradygastria | 66.32
  Par. 2; Day 4; 20 minutes Post-WL; Normal | 19.43
  Par. 2; Day 4; 20 minutes Post-WL; Tachygastria | 11.7
  Par. 2; Day 4; 20 minutes Post-WL; Duodenal | 2.55
  Par. 2; Day 4; 30 minutes Post-WL; Bradygastria | 73.05
  Par. 2; Day 4; 30 minutes Post-WL; Normal | 19.64
  Par. 2; Day 4; 30 minutes Post-WL; Tachygastria | 6.47
  Par. 2; Day 4; 30 minutes Post-WL; Duodenal | 0.84
  Par. 3; Day 1; Pre-WL; Bradygastria | 59.66
  Par. 3; Day 1; Pre-WL; Normal | 9.05
  Par. 3; Day 1; Pre-WL; Tachygastria | 22.39
  Par. 3; Day 1; Pre-WL; Duodenal | 8.91
  Par. 3; Day 1; 10 minutes Post-WL; Bradygastria | 32.73
  Par. 3; Day 1; 10 minutes Post-WL; Normal | 11.03
  Par. 3; Day 1; 10 minutes Post-WL; Tachygastria | 48.77
  Par. 3; Day 1; 10 minutes Post-WL; Duodenal | 7.47
  Par. 3; Day 1; 20 minutes Post-WL; Bradygastria | 29.94
  Par. 3; Day 1; 20 minutes Post-WL; Normal | 22.84
  Par. 3; Day 1; 20 minutes Post-WL; Tachygastria | 39.72
  Par. 3; Day 1; 20 minutes Post-WL; Duodenal | 7.5
  Par. 3; Day 1; 30 minutes Post-WL; Bradygastria | 16.32
  Par. 3; Day 1; 30 minutes Post-WL; Normal | 22.48
  Par. 3; Day 1; 30 minutes Post-WL; Tachygastria | 54.77
  Par. 3; Day 1; 30 minutes Post-WL; Duodenal | 6.43
  Par. 3; Day 4; Pre-WL; Bradygastria | 52.85
  Par. 3; Day 4; Pre-WL; Normal | 16.64
  Par. 3; Day 4; Pre-WL; Tachygastria | 13.21
  Par. 3; Day 4; Pre-WL; Duodenal | 17.29
  Par. 3; Day 4; 10 minutes Post-WL; Bradygastria | 64.27
  Par. 3; Day 4; 10 minutes Post-WL; Normal | 10.37
  Par. 3; Day 4; 10 minutes Post-WL; Tachygastria | 13.26
  Par. 3; Day 4; 10 minutes Post-WL; Duodenal | 12.1
  Par. 3; Day 4; 20 minutes Post-WL; Bradygastria | 71.66
  Par. 3; Day 4; 20 minutes Post-WL; Normal | 11.11
  Par. 3; Day 4; 20 minutes Post-WL; Tachygastria | 9.52
  Par. 3; Day 4; 20 minutes Post-WL; Duodenal | 7.72
  Par. 3; Day 4; 30 minutes Post-WL; Bradygastria | 53.97
  Par. 3; Day 4; 30 minutes Post-WL; Normal | 8.61
  Par. 3; Day 4; 30 minutes Post-WL; Tachygastria | 16.12
  Par. 3; Day 4; 30 minutes Post-WL; Duodenal | 21.3
  Par. 4; Day 1; Pre-WL; Bradygastria | 82.47
  Par. 4; Day 1; Pre-WL; Normal | 6.66
  Par. 4; Day 1; Pre-WL; Tachygastria | 7.86
  Par. 4; Day 1; Pre-WL; Duodenal | 3.01
  Par. 4; Day 1; 10 minutes Post-WL; Bradygastria | 81.89
  Par. 4; Day 1; 10 minutes Post-WL; Normal | 5.6
  Par. 4; Day 1; 10 minutes Post-WL; Tachygastria | 11.63
  Par. 4; Day 1; 10 minutes Post-WL; Duodenal | 0.88
  Par. 4; Day 1; 20 minutes Post-WL; Bradygastria | 62.96
  Par. 4; Day 1; 20 minutes Post-WL; Normal | 12.84
  Par. 4; Day 1; 20 minutes Post-WL; Tachygastria | 17.04
  Par. 4; Day 1; 20 minutes Post-WL; Duodenal | 7.17
  Par. 4; Day 1; 30 minutes Post-WL; Bradygastria | 73.64
  Par. 4; Day 1; 30 minutes Post-WL; Normal | 12.7
  Par. 4; Day 1; 30 minutes Post-WL; Tachygastria | 11.1
  Par. 4; Day 1; 30 minutes Post-WL; Duodenal | 2.56
  Par. 4; Day 4; Pre-WL; Bradygastria | 54.98
  Par. 4; Day 4; Pre-WL; Normal | 17.6
  Par. 4; Day 4; Pre-WL; Tachygastria | 22.97
  Par. 4; Day 4; Pre-WL; Duodenal | 4.45
  Par. 4; Day 4; 10 minutes Post-WL; Bradygastria | 83.7
  Par. 4; Day 4; 10 minutes Post-WL; Normal | 4.2
  Par. 4; Day 4; 10 minutes Post-WL; Tachygastria | 10.69
  Par. 4; Day 4; 10 minutes Post-WL; Duodenal | 1.4
  Par. 4; Day 4; 20 minutes Post-WL; Bradygastria | 82.96
  Par. 4; Day 4; 20 minutes Post-WL; Normal | 5.92
  Par. 4; Day 4; 20 minutes Post-WL; Tachygastria | 10.1
  Par. 4; Day 4; 20 minutes Post-WL; Duodenal | 1.02
  Par. 4; Day 4; 30 minutes Post-WL; Bradygastria | 39.01
  Par. 4; Day 4; 30 minutes Post-WL; Normal | 42.61
  Par. 4; Day 4; 30 minutes Post-WL; Tachygastria | 16.77
  Par. 4; Day 4; 30 minutes Post-WL; Duodenal | 1.62

2. Primary Outcome: Part A: Ratios of Average Power Post- WLT/Pre-WLT by Frequency Region
Description: The effect of exenatide on gastric myoelectrical activity was assessed by EGG using WLT. EGG with WLT is a standardized test to induce gastric distention and measure myoelectrical responses. The gastric myoelectrical activity is generated by the pacemaker interstitial cells at a normal frequency of 3 cycles per minute. The shift of frequency from normal gastric myoelectrical activity to a slower rhythm is bradygastria or faster rhythm is tachygastria. Individual Par. data for ratios of average power post- WLT/pre-WLT in the bradygastria, normal, tachygastria and duodenal range after treatment with exenatide at 10, 20, and 30 minutes post-WL has been presented.
Time Frame: Up to Day 4
Population: Pharmacodynamic Population
Measure: Number; unit: Ratio
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Ratio
  Par. 1; Day 1; 10 minutes Post-WL; Bradygastria | 0
  Par. 1; Day 1; 10 minutes Post-WL; Normal | 0
  Par. 1; Day 1; 10 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 1; 10 minutes Post-WL; Duodenal | 0
  Par. 1; Day 1; 20 minutes Post-WL; Bradygastria | 0
  Par. 1; Day 1; 20 minutes Post-WL; Normal | 0
  Par. 1; Day 1; 20 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 1; 20 minutes Post-WL; Duodenal | 0
  Par. 1; Day 1; 30 minutes Post-WL; Bradygastria | 0
  Par. 1; Day 1; 30 minutes Post-WL; Normal | 0
  Par. 1; Day 1; 30 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 1; 30 minutes Post-WL; Duodenal | 0
  Par. 1; Day 4; 10 minutes Post-WL; Bradygastria | 0
  Par. 1; Day 4; 10 minutes Post-WL; Normal | 0
  Par. 1; Day 4; 10 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 4; 10 minutes Post-WL; Duodenal | 0
  Par. 1; Day 4; 20 minutes Post-WL; Bradygastria | 0
  Par. 1; Day 4; 20 minutes Post-WL; Normal | 0
  Par. 1; Day 4; 20 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 4; 20 minutes Post-WL; Duodenal | 0
  Par. 1; Day 4; 30 minutes Post-WL; Bradygastria | 0
  Par. 1; Day 4; 30 minutes Post-WL; Normal | 0
  Par. 1; Day 4; 30 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 4; 30 minutes Post-WL; Duodenal | 0
  Par. 2; Day 1; 10 minutes Post-WL; Bradygastria | 0.01
  Par. 2; Day 1; 10 minutes Post-WL; Normal | 0
  Par. 2; Day 1; 10 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 1; 10 minutes Post-WL; Duodenal | 0
  Par. 2; Day 1; 20 minutes Post-WL; Bradygastria | 0.04
  Par. 2; Day 1; 20 minutes Post-WL; Normal | 0.04
  Par. 2; Day 1; 20 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 1; 20 minutes Post-WL; Duodenal | 0
  Par. 2; Day 1; 30 minutes Post-WL; Bradygastria | 0.01
  Par. 2; Day 1; 30 minutes Post-WL; Normal | 0.02
  Par. 2; Day 1; 30 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 1; 30 minutes Post-WL; Duodenal | 0
  Par. 2; Day 4; 10 minutes Post-WL; Bradygastria | 0.03
  Par. 2; Day 4; 10 minutes Post-WL; Normal | 0
  Par. 2; Day 4; 10 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 4; 10 minutes Post-WL; Duodenal | 0
  Par. 2; Day 4; 20 minutes Post-WL; Bradygastria | 0.03
  Par. 2; Day 4; 20 minutes Post-WL; Normal | 0.02
  Par. 2; Day 4; 20 minutes Post-WL; Tachygastria | 0.01
  Par. 2; Day 4; 20 minutes Post-WL; Duodenal | 0
  Par. 2; Day 4; 30 minutes Post-WL; Bradygastria | 0.22
  Par. 2; Day 4; 30 minutes Post-WL; Normal | 0.11
  Par. 2; Day 4; 30 minutes Post-WL; Tachygastria | 0.05
  Par. 2; Day 4; 30 minutes Post-WL; Duodenal | 0.01
  Par. 3; Day 1; 10 minutes Post-WL; Bradygastria | 0.13
  Par. 3; Day 1; 10 minutes Post-WL; Normal | 0.29
  Par. 3; Day 1; 10 minutes Post-WL; Tachygastria | 0.52
  Par. 3; Day 1; 10 minutes Post-WL; Duodenal | 0.2
  Par. 3; Day 1; 20 minutes Post-WL; Bradygastria | 0.2
  Par. 3; Day 1; 20 minutes Post-WL; Normal | 0.99
  Par. 3; Day 1; 20 minutes Post-WL; Tachygastria | 0.7
  Par. 3; Day 1; 20 minutes Post-WL; Duodenal | 0.33
  Par. 3; Day 1; 30 minutes Post-WL; Bradygastria | 0.15
  Par. 3; Day 1; 30 minutes Post-WL; Normal | 1.38
  Par. 3; Day 1; 30 minutes Post-WL; Tachygastria | 1.36
  Par. 3; Day 1; 30 minutes Post-WL; Duodenal | 0.4
  Par. 3; Day 4; 10 minutes Post-WL; Bradygastria | 0.16
  Par. 3; Day 4; 10 minutes Post-WL; Normal | 0.08
  Par. 3; Day 4; 10 minutes Post-WL; Tachygastria | 0.13
  Par. 3; Day 4; 10 minutes Post-WL; Duodenal | 0.09
  Par. 3; Day 4; 20 minutes Post-WL; Bradygastria | 0.2
  Par. 3; Day 4; 20 minutes Post-WL; Normal | 0.1
  Par. 3; Day 4; 20 minutes Post-WL; Tachygastria | 0.11
  Par. 3; Day 4; 20 minutes Post-WL; Duodenal | 0.07
  Par. 3; Day 4; 30 minutes Post-WL; Bradygastria | 0.16
  Par. 3; Day 4; 30 minutes Post-WL; Normal | 0.08
  Par. 3; Day 4; 30 minutes Post-WL; Tachygastria | 0.19
  Par. 3; Day 4; 30 minutes Post-WL; Duodenal | 0.19
  Par. 4; Day 1; 10 minutes Post-WL; Bradygastria | 2.6
  Par. 4; Day 1; 10 minutes Post-WL; Normal | 2.21
  Par. 4; Day 1; 10 minutes Post-WL; Tachygastria | 3.88
  Par. 4; Day 1; 10 minutes Post-WL; Duodenal | 0.76
  Par. 4; Day 1; 20 minutes Post-WL; Bradygastria | 0.89
  Par. 4; Day 1; 20 minutes Post-WL; Normal | 2.24
  Par. 4; Day 1; 20 minutes Post-WL; Tachygastria | 2.52
  Par. 4; Day 1; 20 minutes Post-WL; Duodenal | 2.76
  Par. 4; Day 1; 30 minutes Post-WL; Bradygastria | 1.54
  Par. 4; Day 1; 30 minutes Post-WL; Normal | 3.29
  Par. 4; Day 1; 30 minutes Post-WL; Tachygastria | 2.44
  Par. 4; Day 1; 30 minutes Post-WL; Duodenal | 1.47
  Par. 4; Day 4; 10 minutes Post-WL; Bradygastria | 4.7
  Par. 4; Day 4; 10 minutes Post-WL; Normal | 0.74
  Par. 4; Day 4; 10 minutes Post-WL; Tachygastria | 1.44
  Par. 4; Day 4; 10 minutes Post-WL; Duodenal | 0.97
  Par. 4; Day 4; 20 minutes Post-WL; Bradygastria | 10.24
  Par. 4; Day 4; 20 minutes Post-WL; Normal | 2.28
  Par. 4; Day 4; 20 minutes Post-WL; Tachygastria | 2.98
  Par. 4; Day 4; 20 minutes Post-WL; Duodenal | 1.55
  Par. 4; Day 4; 30 minutes Post-WL; Bradygastria | 3.4
  Par. 4; Day 4; 30 minutes Post-WL; Normal | 11.6
  Par. 4; Day 4; 30 minutes Post-WL; Tachygastria | 3.5
  Par. 4; Day 4; 30 minutes Post-WL; Duodenal | 1.74

3. Primary Outcome: Part A: Percentage of Time With the Dominant EGG Frequencies in the Four Frequency Ranges of Bradygastria, Normal, Tachygastria and Duodenal
Description: The effect of exenatide on gastric myoelectrical activity was assessed by EGG using WLT. EGG with WLT is a standardized test to induce gastric distention and measure myoelectrical responses. The gastric myoelectrical activity is generated by the pacemaker interstitial cells at a normal frequency of 3 cycles per minute. The shift of frequency from normal gastric myoelectrical activity to a slower rhythm is bradygastria or faster rhythm is tachygastria. Individual Par. data for dominant EGG frequencies including bradygastria, normal, tachygastria and duodenal at pre-WL and after treatment with exenatide at pre-WL and 10, 20, 30 minutes post-WL has been presented.
Time Frame: Up to Day 4
Population: Pharmacodynamic Population
Measure: Number; unit: Percentage of time
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Percentage of time
  Par. 1; Day 1; Pre-WL; Bradygastria | 80
  Par. 1; Day 1; Pre-WL; Normal | 20
  Par. 1; Day 1; Pre-WL; Tachygastria | 0
  Par. 1; Day 1; Pre-WL; Duodenal | 0
  Par. 1; Day 1; 10 minutes Post-WL; Bradygastria | 100
  Par. 1; Day 1; 10 minutes Post-WL; Normal | 0
  Par. 1; Day 1; 10 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 1; 10 minutes Post-WL; Duodenal | 0
  Par. 1; Day 1; 20 minutes Post-WL; Bradygastria | 100
  Par. 1; Day 1; 20 minutes Post-WL; Normal | 0
  Par. 1; Day 1; 20 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 1; 20 minutes Post-WL; Duodenal | 0
  Par. 1; Day 1; 30 minutes Post-WL; Bradygastria | 50
  Par. 1; Day 1; 30 minutes Post-WL; Normal | 50
  Par. 1; Day 1; 30 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 1; 30 minutes Post-WL; Duodenal | 0
  Par. 1; Day 4; Pre-WL; Bradygastria | 100
  Par. 1; Day 4; Pre-WL; Normal | 0
  Par. 1; Day 4; Pre-WL; Tachygastria | 0
  Par. 1; Day 4; Pre-WL; Duodenal | 0
  Par. 1; Day 4; 10 minutes Post-WL; Bradygastria | 100
  Par. 1; Day 4; 10 minutes Post-WL; Normal | 0
  Par. 1; Day 4; 10 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 4; 10 minutes Post-WL; Duodenal | 0
  Par. 1; Day 4; 20 minutes Post-WL; Bradygastria | 100
  Par. 1; Day 4; 20 minutes Post-WL; Normal | 0
  Par. 1; Day 4; 20 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 4; 20 minutes Post-WL; Duodenal | 0
  Par. 1; Day 4; 30 minutes Post-WL; Bradygastria | 50
  Par. 1; Day 4; 30 minutes Post-WL; Normal | 50
  Par. 1; Day 4; 30 minutes Post-WL; Tachygastria | 0
  Par. 1; Day 4; 30 minutes Post-WL; Duodenal | 0
  Par. 2; Day 1; Pre-WL; Bradygastria | 100
  Par. 2; Day 1; Pre-WL; Normal | 0
  Par. 2; Day 1; Pre-WL; Tachygastria | 0
  Par. 2; Day 1; Pre-WL; Duodenal | 0
  Par. 2; Day 1; 10 minutes Post-WL; Bradygastria | 100
  Par. 2; Day 1; 10 minutes Post-WL; Normal | 0
  Par. 2; Day 1; 10 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 1; 10 minutes Post-WL; Duodenal | 0
  Par. 2; Day 1; 20 minutes Post-WL; Bradygastria | 100
  Par. 2; Day 1; 20 minutes Post-WL; Normal | 0
  Par. 2; Day 1; 20 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 1; 20 minutes Post-WL; Duodenal | 0
  Par. 2; Day 1; 30 minutes Post-WL; Bradygastria | 100
  Par. 2; Day 1; 30 minutes Post-WL; Normal | 0
  Par. 2; Day 1; 30 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 1; 30 minutes Post-WL; Duodenal | 0
  Par. 2; Day 4; Pre-WL; Bradygastria | 100
  Par. 2; Day 4; Pre-WL; Normal | 0
  Par. 2; Day 4; Pre-WL; Tachygastria | 0
  Par. 2; Day 4; Pre-WL; Duodenal | 0
  Par. 2; Day 4; 10 minutes Post-WL; Bradygastria | 100
  Par. 2; Day 4; 10 minutes Post-WL; Normal | 0
  Par. 2; Day 4; 10 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 4; 10 minutes Post-WL; Duodenal | 0
  Par. 2; Day 4; 20 minutes Post-WL; Bradygastria | 100
  Par. 2; Day 4; 20 minutes Post-WL; Normal | 0
  Par. 2; Day 4; 20 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 4; 20 minutes Post-WL; Duodenal | 0
  Par. 2; Day 4; 30 minutes Post-WL; Bradygastria | 50
  Par. 2; Day 4; 30 minutes Post-WL; Normal | 50
  Par. 2; Day 4; 30 minutes Post-WL; Tachygastria | 0
  Par. 2; Day 4; 30 minutes Post-WL; Duodenal | 0
  Par. 3; Day 1; Pre-WL; Bradygastria | 100
  Par. 3; Day 1; Pre-WL; Normal | 0
  Par. 3; Day 1; Pre-WL; Tachygastria | 0
  Par. 3; Day 1; Pre-WL; Duodenal | 0
  Par. 3; Day 1; 10 minutes Post-WL; Bradygastria | 100
  Par. 3; Day 1; 10 minutes Post-WL; Normal | 0
  Par. 3; Day 1; 10 minutes Post-WL; Tachygastria | 0
  Par. 3; Day 1; 10 minutes Post-WL; Duodenal | 0
  Par. 3; Day 1; 20 minutes Post-WL; Bradygastria | 0
  Par. 3; Day 1; 20 minutes Post-WL; Normal | 100
  Par. 3; Day 1; 20 minutes Post-WL; Tachygastria | 0
  Par. 3; Day 1; 20 minutes Post-WL; Duodenal | 0
  Par. 3; Day 1; 30 minutes Post-WL; Bradygastria | 0
  Par. 3; Day 1; 30 minutes Post-WL; Normal | 50
  Par. 3; Day 1; 30 minutes Post-WL; Tachygastria | 50
  Par. 3; Day 1; 30 minutes Post-WL; Duodenal | 0
  Par. 3; Day 4; Pre-WL; Bradygastria | 100
  Par. 3; Day 4; Pre-WL; Normal | 0
  Par. 3; Day 4; Pre-WL; Tachygastria | 0
  Par. 3; Day 4; Pre-WL; Duodenal | 0
  Par. 3; Day 4; 10 minutes Post-WL; Bradygastria | 100
  Par. 3; Day 4; 10 minutes Post-WL; Normal | 0
  Par. 3; Day 4; 10 minutes Post-WL; Tachygastria | 0
  Par. 3; Day 4; 10 minutes Post-WL; Duodenal | 0
  Par. 3; Day 4; 20 minutes Post-WL; Bradygastria | 100
  Par. 3; Day 4; 20 minutes Post-WL; Normal | 0
  Par. 3; Day 4; 20 minutes Post-WL; Tachygastria | 0
  Par. 3; Day 4; 20 minutes Post-WL; Duodenal | 0
  Par. 3; Day 4; 30 minutes Post-WL; Bradygastria | 100
  Par. 3; Day 4; 30 minutes Post-WL; Normal | 0
  Par. 3; Day 4; 30 minutes Post-WL; Tachygastria | 0
  Par. 3; Day 4; 30 minutes Post-WL; Duodenal | 0
  Par. 4; Day 1; Pre-WL; Bradygastria | 100
  Par. 4; Day 1; Pre-WL; Normal | 0
  Par. 4; Day 1; Pre-WL; Tachygastria | 0
  Par. 4; Day 1; Pre-WL; Duodenal | 0
  Par. 4; Day 1; 10 minutes Post-WL; Bradygastria | 100
  Par. 4; Day 1; 10 minutes Post-WL; Normal | 0
  Par. 4; Day 1; 10 minutes Post-WL; Tachygastria | 0
  Par. 4; Day 1; 10 minutes Post-WL; Duodenal | 0
  Par. 4; Day 1; 20 minutes Post-WL; Bradygastria | 100
  Par. 4; Day 1; 20 minutes Post-WL; Normal | 0
  Par. 4; Day 1; 20 minutes Post-WL; Tachygastria | 0
  Par. 4; Day 1; 20 minutes Post-WL; Duodenal | 0
  Par. 4; Day 1; 30 minutes Post-WL; Bradygastria | 100
  Par. 4; Day 1; 30 minutes Post-WL; Normal | 0
  Par. 4; Day 1; 30 minutes Post-WL; Tachygastria | 0
  Par. 4; Day 1; 30 minutes Post-WL; Duodenal | 0
  Par. 4; Day 4; Pre-WL; Bradygastria | 100
  Par. 4; Day 4; Pre-WL; Normal | 0
  Par. 4; Day 4; Pre-WL; Tachygastria | 0
  Par. 4; Day 4; Pre-WL; Duodenal | 0
  Par. 4; Day 4; 10 minutes Post-WL; Bradygastria | 100
  Par. 4; Day 4; 10 minutes Post-WL; Normal | 0
  Par. 4; Day 4; 10 minutes Post-WL; Tachygastria | 0
  Par. 4; Day 4; 10 minutes Post-WL; Duodenal | 0
  Par. 4; Day 4; 20 minutes Post-WL; Bradygastria | 100
  Par. 4; Day 4; 20 minutes Post-WL; Normal | 0
  Par. 4; Day 4; 20 minutes Post-WL; Tachygastria | 0
  Par. 4; Day 4; 20 minutes Post-WL; Duodenal | 0
  Par. 4; Day 4; 30 minutes Post-WL; Bradygastria | 0
  Par. 4; Day 4; 30 minutes Post-WL; Normal | 80
  Par. 4; Day 4; 30 minutes Post-WL; Tachygastria | 20
  Par. 4; Day 4; 30 minutes Post-WL; Duodenal | 0

4. Primary Outcome: Part A: Number of Par. With Shifts in Gastric Rhythm Status
Description: EGG is a technique used to assess gastric myoelectrical activity and thereby gastric rhythm. This analysis was planned as data dependent and not performed as the study was terminated early which resulted in few Par.
Time Frame: Up to 12 days
Population: Pharmacodynamic Population. This analysis was planned as data dependent and not performed as the study was terminated early which resulted in few Par.
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 0

5. Primary Outcome: Part A: Number Par. by Gastric Rhythm Status
Description: as for outcome 4
Time Frame: Up to 12 days
Population: as for outcome 4
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 0

6. Primary Outcome: Part A: Average Dominant Frequency
Description: The effect of exenatide on gastric myoelectrical activity was assessed by EGG using WLT. An EGG with WLT is a standardized test to induce gastric distention and measure myoelectrical responses. The gastric myoelectrical activity is generated by the pacemaker interstitial cells at a normal frequency of 3 cycles per minute. The shift of frequency from normal gastric myoelectrical activity to a slower rhythm is bradygastria or faster rhythm is tachygastria. Individual Par. data for average dominant frequency in the bradygastria, normal, tachygastria and duodenal range after treatment with exenatide at Pre-WL and 10, 20, 30 minutes post-WL has been presented.
Time Frame: Up to Day 4
Population: Pharmacodynamic Population
Measure: Number; unit: Cycles per minute
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Cycles per minute
  Par. 1; Day 1; Pre-WL; Bradygastria | 1.5
  Par. 1; Day 1; 10 minutes Post-WL; Bradygastria | 0.75
  Par. 1; Day 1; 20 minutes Post-WL; Bradygastria | 1.25
  Par. 1; Day 1; 30 minutes Post-WL; Bradygastria | 2.19
  Par. 1; Day 4; Pre-WL; Bradygastria | 1.05
  Par. 1; Day 4; 10 minutes Post-WL; Bradygastria | 0.96
  Par. 1; Day 4; 20 minutes Post-WL; Bradygastria | 1.25
  Par. 1; Day 4; 30 minutes Post-WL; Bradygastria | 2.38
  Par. 2; Day 1; Pre-WL; Bradygastria | 1
  Par. 2; Day 1; 10 minutes Post-WL; Bradygastria | 1
  Par. 2; Day 1; 20 minutes Post-WL; Bradygastria | 1.5
  Par. 2; Day 1; 30 minutes Post-WL; Bradygastria | 1.75
  Par. 2; Day 4; Pre-WL; Bradygastria | 0.75
  Par. 2; Day 4; 10 minutes Post-WL; Bradygastria | 1.38
  Par. 2; Day 4; 20 minutes Post-WL; Bradygastria | 1
  Par. 2; Day 4; 30 minutes Post-WL; Bradygastria | 2.42
  Par. 3; Day 1; Pre-WL; Bradygastria | 0.96
  Par. 3; Day 1; 10 minutes Post-WL; Bradygastria | 1.83
  Par. 3; Day 1; 20 minutes Post-WL; Normal | 3
  Par. 3; Day 1; 30 minutes Post-WL; Tachygastria | 4.13
  Par. 3; Day 4; Pre-WL; Bradygastria | 1.2
  Par. 3; Day 4; 10 minutes Post-WL; Bradygastria | 1.5
  Par. 3; Day 4; 20 minutes Post-WL; Bradygastria | 0.94
  Par. 3; Day 4; 30 minutes Post-WL; Bradygastria | 1.5
  Par. 4; Day 1; Pre-WL; Bradygastria | 0.86
  Par. 4; Day 1; 10 minutes Post-WL; Bradygastria | 1.88
  Par. 4; Day 1; 20 minutes Post-WL; Bradygastria | 1.7
  Par. 4; Day 1; 30 minutes Post-WL; Bradygastria | 1.19
  Par. 4; Day 4; Pre-WL; Bradygastria | 1.2
  Par. 4; Day 4; 10 minutes Post-WL; Bradygastria | 0.94
  Par. 4; Day 4; 20 minutes Post-WL; Bradygastria | 1.29
  Par. 4; Day 4; 30 minutes Post-WL; Normal | 2.9

7. Primary Outcome: Part A: Assessment of Nausea by Visual Analogue Scale (VAS) Score
Description: The effect of exenatide on gastric myoelectrical activity was evaluated using EGG with WLT. An EGG with WLT is a standardized test to induce gastric distention and collect VAS of upper gastrointestinal symptoms. The gastric distention produced by the WL induces nausea in Par. allowing the assessment of gastric myoelectrical activity during the episodes of nausea. The intensity of upper gastrointestinal symptom of nausea was measured using VAS ranging from 0 (no nausea) to 100 (severe nausea) immediately before (pre-WL) and 10, 20, 30 minutes post-WL. Individual Par. responses to VAS score scale has been presented.
Time Frame: Day 4
Population: Pharmacodynamic Population
Measure: Number; unit: Scores on a scale
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Scores on a scale
  Par. 1; Day 4; Pre-WL | 4
  Par. 1; Day 4; 10 minutes Post-WL | 2
  Par. 1; Day 4; 20 minutes Post-WL | 4
  Par. 1; Day 4; 30 minutes Post-WL | 3
  Par. 2; Day 4; Pre-WL | 3
  Par. 2; Day 4; 10 minutes Post-WL | 4
  Par. 2; Day 4; 20 minutes Post-WL | 4
  Par. 2; Day 4; 30 minutes Post-WL | 24
  Par. 3; Day 4; Pre-WL | 1
  Par. 3; Day 4; 10 minutes Post-WL | 0
  Par. 3; Day 4; 20 minutes Post-WL | 0
  Par. 3; Day 4; 30 minutes Post-WL | 0
  Par. 4; Day 4; Pre-WL | 4
  Par. 4; Day 4; 10 minutes Post-WL | 5
  Par. 4; Day 4; 20 minutes Post-WL | 3
  Par. 4; Day 4; 30 minutes Post-WL | 4

8. Primary Outcome: Part A: Time to Half-gastric Emptying
Description: Breath samples were collected to assess the time to half gastric emptying using gastric emptying breath test (GEBT) containing 13 Carbon (13C)-Spirulina pre-meal and post GEBT meal. The GEBT method was used to measure GE of solid food. The time to half gastric emptying for individual Par. has been presented.
Time Frame: Up to Day 5
Population: Pharmacodynamic Population
Measure: Number; unit: Minutes
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Minutes
  Par. 1; Day -1 | 87.2
  Par. 1; Day 5 | 226.5
  Par. 2; Day -1 | 73.0
  Par. 2; Day 5 | 75.5
  Par. 3; Day -1 | 57.6
  Par. 3; Day 5 | 174.0
  Par. 4; Day -1 | 52.9
  Par. 4; Day 5 | 103.8

9. Primary Outcome: Part A: Rate of [13]C Dose Excreted in Breath
Description: The effect of exenatide on gastric emptying was be assessed by calculating the percent dose excreted of 13C in breath multiplied by 1000 (kPCD). Breath samples were collected at the indicated time points. Individual Par. data at pre-meal and 45, 90, 120, 150, 180 and 240 minutes post-meal has been presented.
Time Frame: Day 5
Population: Pharmacodynamic Population
Measure: Number; unit: kPCD per minute
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
kPCD per minute
  Par. 1; Day 5; Pre-Meal | 0
  Par. 1; Day 5; 45 Minutes Post-Meal | 1.8
  Par. 1; Day 5; 90 Minutes Post-Meal | 3.3
  Par. 1; Day 5; 120 Minutes Post-Meal | 3.1
  Par. 1; Day 5; 150 Minutes Post-Meal | 3.3
  Par. 1; Day 5; 180 Minutes Post-Meal | 7.4
  Par. 1; Day 5; 240 Minutes Post-Meal | 21.1
  Par. 2; Day 5; Pre-Meal | 0
  Par. 2; Day 5; 45 Minutes Post-Meal | 22.2
  Par. 2; Day 5; 90 Minutes Post-Meal | 42.5
  Par. 2; Day 5; 120 Minutes Post-Meal | 66.5
  Par. 2; Day 5; 150 Minutes Post-Meal | 82.3
  Par. 2; Day 5; 180 Minutes Post-Meal | 84.7
  Par. 2; Day 5; 240 Minutes Post-Meal | 75.8
  Par. 3; Day 5; Pre-Meal | 0
  Par. 3; Day 5; 45 Minutes Post-Meal | 1
  Par. 3; Day 5; 90 Minutes Post-Meal | 2.3
  Par. 3; Day 5; 120 Minutes Post-Meal | 6.5
  Par. 3; Day 5; 150 Minutes Post-Meal | 16.4
  Par. 3; Day 5; 180 Minutes Post-Meal | 28.2
  Par. 3; Day 5; 240 Minutes Post-Meal | 56.3
  Par. 4; Day 5; Pre-Meal | 0
  Par. 4; Day 5; 45 Minutes Post-Meal | 11.3
  Par. 4; Day 5; 90 Minutes Post-Meal | 27.8
  Par. 4; Day 5; 120 Minutes Post-Meal | 39.6
  Par. 4; Day 5; 150 Minutes Post-Meal | 51.1
  Par. 4; Day 5; 180 Minutes Post-Meal | 59.8
  Par. 4; Day 5; 240 Minutes Post-Meal | 61.6

10. Primary Outcome: Part A: Gastroparesis Cardinal Symptom Index -Daily Diary (GCSI-DD) Score
Description: GCSI-DD is a questionnaire of gastroparesis symptom severity covering the following domains: episodes (epi) of vomiting, epi of retching, nausea/vomiting, fullness/early satiety, and bloating. GCSI-DD contains two symptom severity items upper abdominal pain and overall rating of gastroparesis symptoms. Par. rate each symptom on a 6-point scale from 0 (none), 1 (very mild), 2 (mild), 3 (moderate), 4 (severe),to 5 (very severe). Individual Par. data has been presented. All Subjects Population was used which consisted of all Par. who received at least one dose of study medication.
Time Frame: Up to Day 5
Population: All Subjects Population
Measure: Number; unit: Scores on GCSI-DD scale
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Scores on GCSI-DD scale
  Par. 1; Day-1; Epi of vomiting | 0
  Par. 1; Day 1; Epi of vomiting | 0
  Par. 1; Day 4; Epi of vomiting | 0
  Par. 1; Day 5; Epi of vomiting | 0
  Par. 1; Day -1; Epi of retching | 0
  Par. 1; Day 1; Epi of retching | 0
  Par. 1; Day 4; Epi of retching | 0
  Par. 1; Day 5; Epi of retching | 0
  Par 1; Day -1; Nausea | 0
  Par 1; Day 1; Nausea | 0
  Par 1; Day 4; Nausea | 2
  Par 1; Day 5; Nausea | 1
  Par 1; Day -1; Excessively full after meals | 2
  Par 1; Day 1; Excessively full after meals | 2
  Par 1; Day 4; Excessively full after meals | 5
  Par 1; Day 5; Excessively full after meals | 2
  Par 1; Day -1; Bloating | 0
  Par 1; Day 1; Bloating | 0
  Par 1; Day 4; Bloating | 0
  Par 1; Day 5; Bloating | 5
  Par 1; Day -1; Unable to finish normal-sized meal | 2
  Par 1; Day 1; Unable to finish normal-sized meal | 2
  Par 1; Day 4; Unable to finish normal-sized meal | 5
  Par 1; Day 5; Unable to finish normal-sized meal | 2
  Par 1; Day -1; Retching | 0
  Par 1; Day 1; Retching | 0
  Par 1; Day 4; Retching | 2
  Par 1; Day 5; Retching | 1
  Par 1; Day -1; Vomiting | 0
  Par 1; Day 1; Vomiting | 0
  Par 1; Day 4; Vomiting | 0
  Par 1; Day 5; Vomiting | 0
  Par 1; Day -1; Stomach or belly visibly larger | 0
  Par 1; Day 1; Stomach or belly visibly larger | 0
  Par 1; Day 4; Stomach or belly visibly larger | 0
  Par 1; Day 5; Stomach or belly visibly larger | 0
  Par 1; Day -1; Stomach fullness | 2
  Par 1; Day 1; Stomach fullness | 2
  Par 1; Day 4; Stomach fullness | 5
  Par 1; Day 5; Stomach fullness | 5
  Par 1; Day -1; Loss of appetite | 2
  Par 1; Day 1; Loss of appetite | 2
  Par 1; Day 4; Loss of appetite | 0
  Par 1; Day 5; Loss of appetite | 2
  Par 1; Day -1; Upper abdominal pain | 0
  Par 1; Day 1; Upper abdominal pain | 0
  Par 1; Day 4; Upper abdominal pain | 0
  Par 1; Day 5; Upper abdominal pain | 3
  Par 1; Day -1; Upper abdominal discomfort | 0
  Par 1; Day 1; Upper abdominal discomfort | 0
  Par 1; Day 4; Upper abdominal discomfort | 0
  Par 1; Day 5; Upper abdominal discomfort | 3
  Par 1; Day -1; Overall severity of gastroparesis | 0
  Par 1; Day 1; Overall severity of gastroparesis | 0
  Par 1; Day 4; Overall severity of gastroparesis | 0
  Par 1; Day 5; Overall severity of gastroparesis | 4
  Par. 2; Day -1; Epi of vomiting | 0
  Par. 2; Day 1; Epi of vomiting | 0
  Par. 2; Day 4; Epi of vomiting | 0
  Par. 2; Day 5; Epi of vomiting | 0
  Par. 2; Day -1; Epi of retching | 0
  Par. 2; Day 1; Epi of retching | 0
  Par. 2; Day 4; Epi of retching | 0
  Par. 2; Day 5; Epi of retching | 0
  Par. 2; Day -1; Nausea | 0
  Par. 2 Day 1; Nausea | 0
  Par. 2; Day 4; Nausea | 0
  Par. 2; Day 5; Nausea | 0
  Par. 2; Day -1; Excessively full after meals | 0
  Par. 2; Day 1; Excessively full after meals | 0
  Par. 2; Day 4; Excessively full after meals | 0
  Par. 2; Day 5; Excessively full after meals | 0
  Par. 2; Day -1; Bloating | 0
  Par. 2; Day 1; Bloating | 0
  Par. 2; Day 4; Bloating | 0
  Par. 2; Day 5; Bloating | 0
  Par. 2; Day -1; Unable to finish normal-sized meal | 0
  Par. 2; Day 1; Unable to finish normal-sized meal | 0
  Par. 2; Day 4; Unable to finish normal-sized meal | 0
  Par. 2; Day 5; Unable to finish normal-sized meal | 0
  Par. 2; Day -1; Retching | 0
  Par. 2; Day 1; Retching | 0
  Par. 2; Day 4; Retching | 0
  Par. 2; Day 5; Retching | 0
  Par. 2; Day -1; Vomiting | 0
  Par. 2; Day 1; Vomiting | 0
  Par. 2; Day 4; Vomiting | 0
  Par. 2; Day 5; Vomiting | 0
  Par. 2; Day -1; Stomach or belly visibly larger | 0
  Par. 2; Day 1; Stomach or belly visibly larger | 0
  Par. 2; Day 4; Stomach or belly visibly larger | 0
  Par. 2; Day 5; Stomach or belly visibly larger | 0
  Par. 2; Day -1; Stomach fullness | 0
  Par. 2; Day 1; Stomach fullness | 0
  Par. 2; Day 4; Stomach fullness | 1
  Par. 2; Day 5; Stomach fullness | 0
  Par. 2; Day -1; Loss of appetite | 0
  Par. 2; Day 1; Loss of appetite | 0
  Par. 2; Day 4; Loss of appetite | 0
  Par. 2; Day 5; Loss of appetite | 0
  Par. 2; Day -1; Upper abdominal pain | 0
  Par. 2; Day 1; Upper abdominal pain | 0
  Par. 2; Day 4; Upper abdominal pain | 0
  Par. 2; Day 5; Upper abdominal pain | 0
  Par. 2; Day -1; Upper abdominal discomfort | 0
  Par. 2; Day 1; Upper abdominal discomfort | 0
  Par. 2; Day 4; Upper abdominal discomfort | 0
  Par. 2; Day 5; Upper abdominal discomfort | 0
  Par. 2; Day -1; Overall severity of gastroparesis | 0
  Par. 2; Day 1; Overall severity of gastroparesis | 0
  Par. 2; Day 4; Overall severity of gastroparesis | 0
  Par. 2; Day 5; Overall severity of gastroparesis | 0
  Par. 3; Day -1; Epi of vomiting | 0
  Par. 3; Day 1; Epi of vomiting | 0
  Par. 3; Day 4; Epi of vomiting | 0
  Par. 3; Day 5; Epi of vomiting | 0
  Par. 3; Day -1; Epi of retching | 0
  Par. 3; Day 1; Epi of retching | 0
  Par. 3; Day 4; Epi of retching | 0
  Par. 3; Day 5; Epi of retching | 0
  Par. 3; Day -1; Nausea | 0
  Par. 3; Day 1; Nausea | 0
  Par. 3; Day 4; Nausea | 0
  Par. 3; Day 5; Nausea | 0
  Par. 3; Day -1; Excessively full after meals | 0
  Par. 3; Day 1; Excessively full after meals | 0
  Par. 3; Day 4; Excessively full after meals | 0
  Par. 3; Day 5; Excessively full after meals | 0
  Par. 3; Day -1; Bloating | 0
  Par. 3; Day 1; Bloating | 0
  Par. 3; Day 4; Bloating | 0
  Par. 3; Day 5; Bloating | 0
  Par. 3; Day -1; Unable to finish normal-sized meal | 0
  Par. 3; Day 1; Unable to finish normal-sized meal | 0
  Par. 3; Day 4; Unable to finish normal-sized meal | 0
  Par. 3; Day 5; Unable to finish normal-sized meal | 0
  Par. 3; Day -1; Retching | 0
  Par. 3; Day 1; Retching | 0
  Par. 3; Day 4; Retching | 0
  Par. 3; Day 5; Retching | 0
  Par. 3; Day -1; Vomiting | 0
  Par. 3; Day 1; Vomiting | 0
  Par. 3; Day 4; Vomiting | 0
  Par. 3; Day 5; Vomiting | 0
  Par. 3; Day -1; Stomach or belly visibly larger | 0
  Par. 3; Day 1; Stomach or belly visibly larger | 0
  Par. 3; Day 4; Stomach or belly visibly larger | 0
  Par. 3; Day 5; Stomach or belly visibly larger | 0
  Par. 3; Day -1; Stomach fullness | 0
  Par. 3; Day 1; Stomach fullness | 0
  Par. 3; Day 4; Stomach fullness | 0
  Par. 3; Day 5; Stomach fullness | 0
  Par. 3; Day -1; Loss of appetite | 0
  Par. 3; Day 1; Loss of appetite | 0
  Par. 3; Day 4; Loss of appetite | 0
  Par. 3; Day 5; Loss of appetite | 0
  Par. 3; Day -1; Upper abdominal pain | 0
  Par. 3; Day 1; Upper abdominal pain | 0
  Par. 3; Day 4; Upper abdominal pain | 0
  Par. 3; Day 5; Upper abdominal pain | 0
  Par. 3; Day -1; Upper abdominal discomfort | 0
  Par. 3; Day 1; Upper abdominal discomfort | 0
  Par. 3; Day 4; Upper abdominal discomfort | 0
  Par. 3; Day 5; Upper abdominal discomfort | 0
  Par. 3; Day -1; Overall severity of gastroparesis | 0
  Par. 3; Day 1; Overall severity of gastroparesis | 0
  Par. 3; Day 4; Overall severity of gastroparesis | 0
  Par. 3; Day 5; Overall severity of gastroparesis | 0
  Par. 4; Day -1; Epi of vomiting | 0
  Par. 4; Day 1; Epi of vomiting | 0
  Par. 4; Day 4; Epi of vomiting | 0
  Par. 4; Day 5; Epi of vomiting | 0
  Par. 4; Day -1; Epi of retching | 0
  Par. 4; Day 1; Epi of retching | 0
  Par. 4; Day 4; Epi of retching | 0
  Par. 4; Day 5; Epi of retching | 0
  Par. 4; Day -1; Nausea | 0
  Par. 4; Day 1; Nausea | 0
  Par. 4; Day 4; Nausea | 0
  Par. 4; Day 5; Nausea | 0
  Par. 4; Day -1; Excessively full after meals | 0
  Par. 4; Day 1; Excessively full after meals | 1
  Par. 4; Day 4; Excessively full after meals | 1
  Par. 4; Day 5; Excessively full after meals | 0
  Par. 4; Day -1; Bloating | 0
  Par. 4; Day 1; Bloating | 1
  Par. 4; Day 4; Bloating | 0
  Par. 4; Day 5; Bloating | 0
  Par.4; Day -1; Unable to finish normal-sized meal | 0
  Par.4; Day 1; Unable to finish normal-sized meal | 0
  Par.4; Day 4; Unable to finish normal-sized meal | 0
  Par.4; Day 5; Unable to finish normal-sized meal | 0
  Par. 4; Day -1; Retching | 0
  Par. 4; Day 1; Retching | 0
  Par. 4; Day 4; Retching | 0
  Par. 4; Day 5; Retching | 0
  Par. 4; Day -1; Vomiting | 0
  Par. 4; Day 1; Vomiting | 0
  Par. 4; Day 4; Vomiting | 0
  Par. 4; Day 5; Vomiting | 0
  Par. 4; Day -1; Stomach or belly visibly larger | 0
  Par. 4; Day 1; Stomach or belly visibly larger | 0
  Par. 4; Day 4; Stomach or belly visibly larger | 0
  Par. 4; Day 5; Stomach or belly visibly larger | 0
  Par. 4; Day -1; Stomach fullness | 0
  Par. 4; Day 1; Stomach fullness | 1
  Par. 4; Day 4; Stomach fullness | 1
  Par. 4; Day 5; Stomach fullness | 0
  Par. 4; Day -1; Loss of appetite | 0
  Par. 4; Day 1; Loss of appetite | 0
  Par. 4; Day 4; Loss of appetite | 0
  Par. 4; Day 5; Loss of appetite | 0
  Par. 4; Day -1; Upper abdominal pain | 0
  Par. 4; Day 1; Upper abdominal pain | 0
  Par. 4; Day 4; Upper abdominal pain | 0
  Par. 4; Day 5; Upper abdominal pain | 0
  Par. 4; Day -1; Upper abdominal discomfort | 0
  Par. 4; Day 1; Upper abdominal discomfort | 0
  Par. 4; Day 4; Upper abdominal discomfort | 0
  Par. 4; Day 5; Upper abdominal discomfort | 0
  Par. 4; Day -1; Overall severity of gastroparesis | 0
  Par. 4; Day 1; Overall severity of gastroparesis | 1
  Par. 4; Day 4; Overall severity of gastroparesis | 1
  Par. 4; Day 5; Overall severity of gastroparesis | 0

11. Primary Outcome: Part A: The Volume of Water Ingested During EGG
Description: The volume of water consumed by Par. at indicated time points after treatment with exenatide during EGG with WLT was determined. An EGG with WLT is a standardized test to induce gastric distention. Individual Par. data has been presented.
Time Frame: Up to Day 4
Population: Pharmacodynamic Population
Measure: Number; unit: Milliliter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Milliliter
  Par. 1; Day 1 | 430
  Par. 1; Day 4 | 360
  Par. 2; Day 1 | 2160
  Par. 2; Day 4 | 1980
  Par. 3; Day 1 | 900
  Par. 3; Day 4 | 1080
  Par. 4; Day 1 | 1000
  Par. 4; Day 4 | 1000

12. Primary Outcome: Part A: Assessment of Stomach Fullness, Hunger, Bloating and Abdominal Pain by VAS Score
Description: The effect of exenatide on gastric myoelectrical activity was evaluated using EGG with WLT. An EGG with WLT is a standardized test to induce gastric distention and collect VAS of upper gastrointestinal symptoms. The gastric distention produced by the WL induces upper gastrointestinal symptoms including stomach fullness, hunger, bloating and abdominal pain in Par. allowing the assessment of gastric myoelectrical activity. The intensity of upper gastrointestinal symptoms was measured using VAS scores ranging from stomach empty (0) to stomach full (100), hunger (0) to satiety (100) and no bloating (0) to severe bloating (100). Individual Par. responses to VAS has been presented.
Time Frame: Day 4
Population: Pharmacodynamic Population
Measure: Number; unit: Scores on VAS scale
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Scores on VAS scale
  Par. 1; Day 4; Pre-WL; Stomach fullness | 3
  Par. 1; Day 4; 10 minutes Post-WL;Stomach fullness | 43
  Par. 1; Stomach fullness;Day 4; 20 minutes Post-WL | 50
  Par. 1; Day 4; 30 minutes Post-WL;Stomach fullness | 9
  Par. 2; Day 4; Pre-WL;Stomach fullness | 11
  Par. 2; Day 4; 10 minutes Post-WL;Stomach fullness | 94
  Par. 2; Day 4; 20 minutes Post-WL;Stomach fullness | 92
  Par. 2; Day 4; 30 minutes Post-WL;Stomach fullness | 85
  Par. 3; Day 4; Pre-WL; Stomach fullness | 10
  Par. 3; Day 4; 10 minutes Post-WL;Stomach fullness | 89
  Par. 3; Day 4; 20 minutes Post-WL;Stomach fullness | 82
  Par. 3; Day 4; 30 minutes Post-WL;Stomach fullness | 75
  Par. 4; Day 4; Pre-WL;Stomach fullness | 28
  Par. 4; Day 4; 10 minutes Post-WL;Stomach fullness | 34
  Par. 4; Day 4; 20 minutes Post-WL;Stomach fullness | 38
  Par. 4; Day 4; 30 minutes Post-WL;Stomach fullness | 35
  Par. 1; Day 4; Pre-WL; Bloating | 4
  Par. 1; Day 4; 10 minutes Post-WL;Bloating | 27
  Par. 1; Day 4; 20 minutes Post-WL;Bloating | 46
  Par. 1; Day 4; 30 minutes Post-WL; Bloating | 45
  Par. 2; Day 4; Pre-WL;Bloating | 3
  Par. 2; Day 4; 10 minutes Post-WL;Bloating | 5
  Par. 2; Day 4; 20 minutes Post-WL;Bloating | 6
  Par. 2; Day 4; 30 minutes Post-WL;Bloating | 26
  Par. 3; Bloating; Day 4; Pre-WL;Bloating | 1
  Par. 3; Day 4; 10 minutes Post-WL;Bloating | 0
  Par. 3; Day 4; 20 minutes Post-WL;Bloating | 0
  Par. 3; Day 4; 30 minutes Post-WL;Bloating | 1
  Par. 4; Day 4; Pre-WL; Bloating | 3
  Par. 4; Day 4; 10 minutes Post-WL;Bloating | 22
  Par. 4; Day 4; 20 minutes Post-WL; Bloating | 42
  Par. 4; Bloating; Day 4; 30 minutes Post-WL | 35
  Par. 1; Day 4; Pre-WL; Abdominal pain | 3
  Par. 1; Day 4; 10 minutes Post-WL; Abdominal pain | 4
  Par. 1; Day 4; 20 minutes Post-WL; Abdominal pain | 3
  Par. 1; Day 4; 30 minutes Post-WL;Abdominal pain | 3
  Par. 2; Day 4; Pre-WL; Abdominal pain | 4
  Par. 2; Day 4; 10 minutes Post-WL; Abdominal pain | 4
  Par. 2; Day 4; 20 minutes Post-WL; Abdominal pain | 7
  Par. 2; Day 4; 30 minutes Post-WL;Abdominal pain | 6
  Par. 3; Day 4; Pre-WL; Abdominal pain | 0
  Par. 3;Day 4; 10 minutes Post-WL; Abdominal pain | 0
  Par. 3; Day 4; 20 minutes Post-WL; Abdominal pain | 0
  Par. 3; Day 4; 30 minutes Post-WL; Abdominal pain | 0
  Par. 4; Day 4; Pre-WL; Abdominal pain | 4
  Par. 4; Day 4; 10 minutes Post-WL;Abdominal pain | 4
  Par. 4; Day 4; 20 minutes Post-WL; Abdominal pain | 5
  Par. 4; Day 4; 30 minutes Post-WL; Abdominal pain | 5
  Par. 1; Day 4; Pre-WL; Hunger | 88
  Par. 1; Day 4; 10 minutes Post-WL; Hunger | 79
  Par. 1; Day 4; 20 minutes Post-WL;Hunger | 85
  Par. 1;Day 4; 30 minutes Post-WL;Hunger | 84
  Par. 2; Day 4; Pre-WL;Hunger | 32
  Par. 2; Day 4; 10 minutes Post-WL; Hunger | 16
  Par. 2; Day 4; 20 minutes Post-WL; Hunger | 19
  Par. 2; Day 4; 30 minutes Post-WL; Hunger | 27
  Par. 3; Day 4; Pre-WL; Hunger | 21
  Par. 3; Day 4; 10 minutes Post-WL; Hunger | 3
  Par. 3; Day 4; 20 minutes Post-WL; Hunger | 6
  Par. 3; Day 4; 30 minutes Post-WL;Hunger | 17
  Par. 4; Day 4; Pre-WL;Hunger | 19
  Par. 4; Day 4; 10 minutes Post-WL; Hunger | 16
  Par. 4; Day 4; 20 minutes Post-WL; Hunger | 29
  Par. 4; Day 4; 30 minutes Post-WL;Hunger | 37

13. Primary Outcome: Part A: Assessment of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) as a Measure of Safety
Description: SBP and DBP was measured either in a semi-recumbent or seated position after at least a 5-minute rest period. Individual Par. data for SBP and DBP up to follow-up (up to 12 days) has been presented.
Time Frame: Up to 12 days
Population: All Subjects Population
Measure: Number; unit: Millimeter of mercury
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Millimeter of mercury
  Par. 1; Day -1; SBP | 126
  Par. 1; Day 1; SBP | 121
  Par. 1; Day 4; SBP | 124
  Par. 1; Day 5; SBP | 112
  Par. 1; Follow-up; SBP | 125
  Par. 1; Day -1; DBP | 71
  Par. 1; Day 1; DBP | 61
  Par. 1; Day 4; DBP | 69
  Par. 1; Day 5; DBP | 67
  Par. 1; Follow-up; DBP | 72
  Par. 2; Day -1; SBP | 105
  Par. 2; Day 1; SBP | 109
  Par. 2; Day 4; SBP | 119
  Par. 2; Day 5; SBP | 121
  Par. 2; Follow-up; SBP | 124
  Par. 2; Day -1; DBP | 61
  Par. 2; Day 1; DBP | 68
  Par. 2; Day 4; DBP | 71
  Par. 2; Day 5; DBP | 68
  Par. 2; Follow-up; DBP | 75
  Par. 3; Day -1; SBP | 131
  Par. 3; Day 1; SBP | 131
  Par. 3; Day 4; SBP | 132
  Par. 3; Day 5; SBP | 112
  Par. 3; Follow-up; SBP | 126
  Par. 3; Day -1; DBP | 86
  Par. 3; Day 1; DBP | 82
  Par. 3; Day 4; DBP | 87
  Par. 3; Day 5; DBP | 76
  Par. 3; Follow-up; DBP | 87
  Par. 4; Day -1; SBP | 138
  Par. 4; Day 1; SBP | 139
  Par. 4; Day 4; SBP | 127
  Par. 4; Day 5; SBP | 123
  Par. 4; Follow-up; SBP | 160
  Par. 4; Day -1; DBP | 83
  Par. 4; Day 1; DBP | 90
  Par. 4; Day 4; DBP | 83
  Par. 4; Day 5; DBP | 81
  Par. 4; Follow-up; DBP | 86

14. Primary Outcome: Part A: Assessment of Heart Rate (HR) as a Measure of Safety
Description: HR was measured either in a semi-recumbent or seated position after at least a 5-minute rest period. Individual Par. data for HR up to follow-up (up to 12 days) has been presented.
Time Frame: Up to 12 days
Population: All Subjects Population
Measure: Number; unit: Beats per minute
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Beats per minute
  Par. 1; Day -1 | 69
  Par. 1; Day 1 | 65
  Par. 1; Day 4 | 66
  Par. 1; Day 5 | 84
  Par. 1; Follow-up | 68
  Par. 2; Day -1 | 57
  Par. 2; Day 1 | 64
  Par. 2; Day 4 | 62
  Par. 2; Day 5 | 82
  Par. 2; Follow-up | 58
  Par. 3; Day -1 | 72
  Par. 3; Day 1 | 74
  Par. 3; Day 4 | 78
  Par. 3; Day 5 | 82
  Par. 3; Follow-up | 78
  Par. 4; Day -1 | 78
  Par. 4; Day 1 | 89
  Par. 4; Day 4 | 77
  Par. 4; Day 5 | 82
  Par. 4; Follow-up | 72

15. Primary Outcome: Part A: Basophils, Eosinophil, Lymphocytes, Monocytes, Platelet Count, Total Neutrophils, White Blood Cell (WBC) Level at Indicated Time Points
Description: Blood samples were collected for analysis of hematology parameters including basophils, eosinophil, lymphocytes, monocytes, platelet count, total neutrophils, and WBC. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Giga unit per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Giga unit per liter
  Par.1; Basophils | 0.02
  Par.1; Eosinophils | 0.11
  Par.1; Lymphocytes | 1.57
  Par.1; Monocytes | 0.35
  Par.1; Platelet count | 268
  Par.1; Total Neutrophils | 6.33
  Par.1; WBC | 8.4
  Par.2; Basophils | 0.02
  Par.2; Eosinophils | 0.04
  Par.2; Lymphocytes | 1.39
  Par.2; Monocytes | 0.25
  Par.2; Platelet count | 217
  Par.2; Total Neutrophils | 2.54
  Par.2; WBC | 4.2
  Par.3; Basophils | 0.03
  Par.3; Eosinophils | 0.21
  Par.3; Lymphocytes | 1.77
  Par.3; Monocytes | 0.58
  Par.3; Platelet count | 202
  Par.3; Total Neutrophils | 5.09
  Par.3; WBC | 7.7
  Par.4; Basophils | 0.04
  Par.4; Eosinophils | 0.23
  Par.4; Lymphocytes | 3.06
  Par.4; Monocytes | 0.89
  Par.4; Platelet count | 230
  Par.4; Total Neutrophils | 1.2
  Par.4; WBC | 5.4

16. Primary Outcome: Part A: Red Blood Cell (RBC) Count at Indicated Time Points
Description: Blood samples were collected for analysis of RBC count. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Tetra unit per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Tetra unit per liter
  Par. 1 | 4.7
  Par. 2 | 4.8
  Par. 3 | 5
  Par. 4 | 4.9

17. Primary Outcome: Part A: Hemoglobin Level at Indicated Time Points
Description: Blood samples were collected for analysis of hemoglobin level. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Grams per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Grams per liter
  Par. 1 | 125
  Par. 2 | 133
  Par. 3 | 149
  Par. 4 | 156

18. Primary Outcome: Part A: Hematocrit Level at Indicated Time Points
Description: Blood samples were collected for analysis of hematocrit level. Individual Par. data at indicated time points has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Proportion of RBC in blood
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Proportion of RBC in blood
  Par. 1 | 0.399
  Par. 2 | 0.426
  Par. 3 | 0.466
  Par. 4 | 0.462

19. Primary Outcome: Part A: Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Gamma Glutamyl Transferase (GGT) Levels at Indicated Time Points
Description: Blood samples were collected for analysis of clinical chemistry parameters including ALT, AST and GGT. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: International unit per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
International unit per liter
  Par. 1; ALT | 21
  Par. 1; AST | 20
  Par. 1; GGT | 46
  Par. 2; ALT | 25
  Par. 2; AST | 18
  Par. 2; GGT | 76
  Par. 3; ALT | 11
  Par. 3; AST | 12
  Par. 3; GGT | 19
  Par. 4; ALT | 17
  Par. 4; AST | 20
  Par. 4; GGT | 30

20. Primary Outcome: Part A: Glucose, Calcium, Magnesium, Potassium, Sodium, Phosphorus Inorganic, Chloride, Urea/Blood Urea Nitrogen (BUN) Levels
Description: Blood samples were collected for analysis of glucose, calcium, magnesium, potassium, sodium, phosphorus inorganic, chloride, and urea/BUN levels. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Millimoles per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Millimoles per liter
  Par. 1; Glucose | 9.2
  Par. 1; Calcium | 2.44
  Par. 1; Magnesium | 0.86
  Par. 1; Potassium | 5.6
  Par. 1; Sodium | 139
  Par. 1; Phosphorus inorganic | 1.5
  Par. 1; Chloride | 105
  Par. 1; Urea/BUN | 7.5
  Par. 2; Glucose | 7.5
  Par. 2; Calcium | 2.44
  Par. 2; Magnesium | 0.9
  Par. 2; Potassium | 5.1
  Par. 2; Sodium | 139
  Par. 2; Phosphorus inorganic | 1.25
  Par. 2; Chloride | 105
  Par. 2; Urea/BUN | 6.5
  Par. 3; Glucose | 9.1
  Par. 3; Calcium | 2.38
  Par. 3; Magnesium | 0.8
  Par. 3; Potassium | 4.2
  Par. 3; Sodium | 140
  Par. 3; Phosphorus inorganic | 1.2
  Par. 3; Chloride | 103
  Par. 3; Urea/BUN | 7
  Par. 4; Glucose | 7.9
  Par. 4; Calcium | 2.4
  Par. 4; Magnesium | 0.8
  Par. 4; Potassium | 4.3
  Par. 4; Sodium | 138
  Par. 4; Phosphorus inorganic | 1.15
  Par. 4; Chloride | 101
  Par. 4; Urea/BUN | 4.5

21. Primary Outcome: Part A: Creatinine, Direct Bilirubin, Total Bilirubin, Indirect Bilirubin Levels at Indicated Time Points
Description: Blood samples were collected for analysis of clinical chemistry parameters including creatinine, direct bilirubin, total bilirubin, indirect bilirubin levels. Individual Par. data at indicated time points has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Micromoles per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Micromoles per liter
  Par. 1; Creatinine | 67.2
  Par. 1; Direct Bilirubin | 2
  Par. 1; Total Bilirubin | 10
  Par. 1; Indirect Bilirubin | 8
  Par. 2; Creatinine | 105.2
  Par. 2; Direct Bilirubin | 2
  Par. 2; Total Bilirubin | 6
  Par. 2; Indirect Bilirubin | 4
  Par. 3; Creatinine | 76.9
  Par. 3; Direct Bilirubin | 4
  Par. 3; Total Bilirubin | 16
  Par. 3; Indirect Bilirubin | 12
  Par. 4; Creatinine | 83.1
  Par. 4; Direct Bilirubin | 2
  Par. 4; Total Bilirubin | 6
  Par. 4; Indirect Bilirubin | 4

22. Primary Outcome: Part A: Estimated Glomerular Filtration Rate at Indicated Time Points
Description: Estimated glomerular filtration rate was calculated using the "modification of diet in renal disease" (MDRD) formula by multiplying 175 with serum creatinine^-1.154 multiplied by age^-0.203 multiplied by 0.742 (if female) multiplied by 1.212 (if African American Par.). Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Milliliter per second per 1.73 meter ^2
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Milliliter per second per 1.73 meter ^2
  Part. 1 | 1.3026
  Part. 2 | 1.2859
  Part. 3 | 1.5197
  Part. 4 | 1.6533

23. Primary Outcome: Part A: Total Protein, Albumin Levels at Indicated Time Points
Description: Blood samples were collected for analysis of clinical chemistry parameters including total protein and albumin levels. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Grams per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Grams per liter
  Par. 1; Total Protein | 77
  Par. 1; Albumin levels | 43
  Par. 2; Total Protein | 75
  Par. 2; Albumin levels | 46
  Par. 3; Total Protein | 71
  Par. 3; Albumin levels | 44
  Par. 4; Total Protein | 74
  Par. 4; Albumin levels | 46

24. Primary Outcome: Part A: Albumin Level in Urine at Indicated Time Points
Description: Samples were collected to analyze albumin level in urine. Individual Par. data at indicated time point has been collected.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Milligrams per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Milligrams per liter
  Par. 1 | 35
  Par. 2 | 35
  Par. 3 | 5
  Par. 4 | 5

25. Primary Outcome: Part A: Concentration of Creatinine in Urine at Indicated Time Points
Description: Samples were collected to analyze concentration of creatinine in urine. Individual Par. at indicated time point has been presented at indicated time points.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Micromoles per liter
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Micromoles per liter
  Par. 1 | 12450
  Par. 2 | 16240
  Par. 3 | 13300
  Par. 4 | 22020

26. Primary Outcome: Part A: Number of Par. With Presence of Ketones, Occult Blood, Glucose, Nitrates and Leukocyte Esterase in Urine at Indicated Time Points
Description: Urine samples were collected to analyze presence of ketones, occult blood, glucose, nitrates and leukocyte esterase in urine. The dipstick test gives results in a semi-quantitative manner. NA represents data was not available due to lab data transfer error. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Participants
  Par. 1; Ketones; Negative | 1
  Par 1; Occult blood; Trace | 1
  Par 1; Glucose | NA — NA represents data was not available due to lab data transfer error.
  Par 1; Nitrates | NA — NA represents data was not available due to lab data transfer error.
  Par 1; Leukocyte esterase | NA — NA represents data was not available due to lab data transfer error.
  Par. 2; Ketones; Negative | 1
  Par. 2; Occult blood; Negative | 1
  Par. 2; Glucose | NA — NA represents data was not available due to lab data transfer error.
  Par 2; Nitrates | NA — NA represents data was not available due to lab data transfer error.
  Par 2; Leukocyte esterase | NA — NA represents data was not available due to lab data transfer error.
  Par. 3; Ketones; Negative | 1
  Par. 3; Occult blood; Negative | 1
  Par. 3; Glucose | NA — NA represents data was not available due to lab data transfer error.
  Par 3; Nitrates | NA — NA represents data was not available due to lab data transfer error.
  Par 3; Leukocyte esterase | NA — NA represents data was not available due to lab data transfer error.
  Par. 4; Ketones; Negative | 1
  Par. 4; Occult blood; Negative | 1
  Par. 4; Glucose | NA — NA represents data was not available due to lab data transfer error.
  Par 4; Nitrates | NA — NA represents data was not available due to lab data transfer error.
  Par 4; Leukocyte esterase | NA — NA represents data was not available due to lab data transfer error.

27. Primary Outcome: Part A: Presence RBC and WBC in Urine Assessed by Microscopy
Description: Samples were collected to analyze the presence of RBC and WBC in urine by microscopy. Individual Par. data at indicated time point has been presented. "NA" indicates data was not available as RBC and WBC count would only available if blood or protein were abnormal. The RBC and WBC values of "1" for participant 1 actually reflect 0-1.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: High Power field
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
High Power field
  Par.1; RBC | 1
  Par. 1; WBC | 1
  Par. 2; RBC | NA — NA indicates data was not available as RBC and WBC count would only available if blood or protein were abnormal.
  Par. 2; WBC | NA — NA indicates data was not available as RBC and WBC count would only available if blood or protein were abnormal.
  Par. 3; RBC | NA — NA indicated data was not available as RBC and WBC count would only available if blood or protein were abnormal.
  Part. 3; WBC | NA — NA indicated data was not available as RBC and WBC count would only available if blood or protein were abnormal.
  Part 4; RBC | NA — NA indicated data was not available as RBC and WBC count would only available if blood or protein were abnormal.
  Part. 4; WBC | NA — NA indicated data was not available as RBC and WBC count would only available if blood or protein were abnormal.

28. Primary Outcome: Part A: Specific Gravity of Urine at Indicated Time Points
Description: Urine samples were collected to analyze specific gravity of urine. Specific gravity, is a measure of urine concentration and is measured using a chemical test. Specific gravity measurements provide a comparison of the amount of substances dissolved in urine as compared to pure water. If there were no solutes present, the specific gravity of urine would be 1.000 the same as pure water. Specific gravity between 1.002 and 1.035 could be considered as normal. Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Kilograms per meter^3
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Kilograms per meter^3
  Par. 1 | 1.021
  Par. 2 | 1.019
  Par. 3 | 1.023
  Par. 4 | 1.027

29. Primary Outcome: Part A: Potential of Hydrogen (pH) of Urine at Indicated Time Points
Description: Urine Samples were collected to analyze pH. pH is a measure of hydrogen ion concentration and used to determine the acidity or alkalinity of urine. pH scale ranges from 0 to 14. A neutral pH is 7.0. The higher number indicates the more basic (alkaline) nature of urine and lower the number indicates the more acidic urine.Individual Par. data at indicated time point has been presented.
Time Frame: Day 5
Population: All Subjects Population
Measure: Number; unit: Points on a scale
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Points on a scale
  Par. 1 | 5
  Par. 2 | 5.5
  Par. 3 | 6
  Par. 4 | 5

30. Primary Outcome: Part A: Number of Par. With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation Par. temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function. Number of Par. with AEs and SAEs have been presented.
Time Frame: Up to 12 days
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Participants
  Any AE | 1
  Any SAE | 0

31. Primary Outcome: Part A: Number of Par. With Nausea AEs Presenting Outside the Timing of the WLT and GCSI-DD
Description: GCSI-DD is a questionnaire of gastroparesis symptom severity covering the following domains: nausea/vomiting, fullness/early satiety, and bloating. The effect of exenatide on gastric myoelectrical activity was assessed by EGG using WLT.
Time Frame: Up to 12 days
Population: All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Part A: Exenatide SC Injection
Number analyzed (Participants) | 4
Participants | 0

32. Primary Outcome: Part B: Distribution of Average Power by Frequency Region
Description: EGG is a technique used to assess gastric myoelectrical activity using WLT. An EGG with WLT is a standardized test to induce gastric distention and measure myoelectrical responses. The gastric myoelectrical activity is generated by the pacemaker interstitial cells at a normal frequency of 3 cycles per minute. The shift of frequency from normal gastric myoelectrical activity to a slower rhythm is bradygastria or faster rhythm is tachygastria. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: Pharmacodynamic Population. The data were not collected for Part B because no Par. were enrolled into this part of the study.
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: Part B: Ratios of Average Power Post- WLT/Pre-WLT by Frequency Region
Description: as for outcome 32
Time Frame: Up to 8 weeks
Population: as for outcome 32
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

34. Primary Outcome: Part B: Percentage of Time With the Dominant EGG Frequencies in the Four Frequency Ranges of Bradygastria, Normal, Tachygastria and Duodenal
Description: EGG is a technique used to assess gastric myoelectrical activity using WLT. An EGG with An WLT is a standardized test to induce gastric distention and measure myoelectrical responses. The gastric myoelectrical activity is generated by the pacemaker interstitial cells at a normal frequency of 3 cycles per minute. The shift of frequency from normal gastric myoelectrical activity to a slower rhythm is bradygastria or faster rhythm is tachygastria. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 32
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

35. Primary Outcome: Part B: Assessment of Nausea by VAS Score
Description: The VAS was used to measure the intensity of nausea analyzed on the basis of scores ranging from 0 (no nausea) to 100 (severe nausea). This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 32
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Part B: Time to Half-gastric Emptying
Description: The GEBT containing 13C-Spirulina was used to measure the time to half-gastric emptying. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 32
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Part B: Rate of [13]C Dose Excreted in Breath
Description: The rate of [13]C dose excreted in breath was assessed to study gastric empting using GEBT. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 32
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Part B: The Volume of Water Ingested During EGG
Description: EGG with WLT is a standardized test to induce gastric distention. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 32
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Part B: Assessment of Stomach Fullness, Hunger, Bloating and Abdominal Pain by VAS Score
Description: EGG with WLT is a standardized test to induce gastric distention and collect VAS of upper gastrointestinal symptoms ranging from stomach empty (0) to stomach full (100), hunger (0) to satiety (100) and no bloating (0) to severe bloating (100). The gastric distention produced by the WL induces upper gastrointestinal symptoms including stomach fullness, hunger, bloating and abdominal pain in Par. allowing the assessment of gastric myoelectrical activity. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 32
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Part B: Number of Par. With Abnormal Values for Vital Signs
Description: Vital signs included SBP, DBP and heart rate. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 12 weeks
Population: All Subjects Population. The data were not collected for Part B because no Par. were enrolled into this part of the study.
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Part B: Number of Par. With Abnormal Values for Hematology Parameters
Description: Hematology parameters included basophils, eosinophils, lymphocytes, monocytes, platelet count, total neutrophils, WBC, RBC, hemoglobin and hematocrit levels. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 40
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Part B: Number of Par. With Abnormal Values for Clinical Chemistry Parameters
Description: Clinical chemistry parameters included ALT, AST, GGT, glucose, calcium, magnesium, potassium, sodium, phosphorus inorganic, chloride, BUN, creatinine, direct bilirubin, total bilirubin, indirect bilirubin, glomerular filtration rate (MDRD Enzymatic level), total protein, and albumin level. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 40
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Part B: Number of Par. With Abnormal Values for Urinalysis
Description: Urinalysis included analysis of concentration of creatinine, presence of ketones and occult blood in urine (using dipstick test), presence RBC and WBC in urine (using microscopy), specific gravity and pH of urine. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 40
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Part B: Number of Par. With AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation Par., temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 12 weeks
Population: as for outcome 40
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Part B: Assessment of GCSI-DD Score
Description: GCSI-DD is a questionnaire of gastroparesis symptom severity covering the following domains: nausea/vomiting, fullness/early satiety, and bloating. GCSI-DD contains two symptom severity items upper abdominal pain and overall rating of gastroparesis symptoms. Par. rate each symptom on a 6-point scale from 0 (none), 1 (very mild), 2 (mild), 3 (moderate), 4 (severe) to 5 (very severe). This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 8 weeks
Population: as for outcome 40
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Part B: Number of Par. With Nausea AEs Presenting Outside the Timing of the WLT and GCSI-DD
Description: GCSI-DD is a questionnaire of gastroparesis symptom severity covering the following domains: nausea/vomiting, fullness/early satiety, and bloating. The effect of exenatide on gastric myoelectrical activity was assessed by EGG using WLT. This analysis was planned but not performed for Part B as the study was terminated during Part A.
Time Frame: Up to 12 weeks
Population: as for outcome 40
Arm/Group | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs) and serious adverse events (SAEs) were collected from the start of the study treatment until the follow up (up to 12 days).
Description: AEs and SAEs were collected in Part A from All Subjects Population comprised all Par. who received at least one dose of study medication. The data were not collected for Part B because no Par. were enrolled into this part of the study.
Arm/Group | Part A: Exenatide SC Injection | Part B: Exenatide SC Injection | Part B: Albiglutide SC Injection
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/4 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Exenatide SC Injection (N=4) | Part B: Exenatide SC Injection (N=0) | Part B: Albiglutide SC Injection (N=0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 | 0
Early satiety (General disorders) | 1 (1) | 0 | 0
Feeling jittery (General disorders) | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT02793154/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02793154/SAP_001.pdf